CLINICAL TRIAL: NCT01464801
Title: Long-term Investigation of Resveratrol on Management of Metabolic Syndrome, Osteoporosis and Inflammation, and Identification of Plant Derived Anti-inflammatory Compounds, Study 3
Brief Title: Resveratrol in Patients With Non-alcoholic Fatty Liver Disease
Acronym: LIRMOI3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIRMOI 3
Record Dates: First submitted 2011-09-29; First posted 2011-11-04 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2013-08

CONDITIONS: Fatty Liver
Keywords: Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Resveratrol; Human study
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Experimental): Subjects are given resveratrol 500 mg 3 times daily for 6 months.
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Subjects are given Placebo tablets 3 times daily for 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Tablet Resveratrol 500 mg 3 times daily for 6 months
  Arms: Resveratrol
Dietary Supplement: Placebo — Tablet Placebo 3 times daily for 6 months
  Arms: Placebo

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) and fatty liver hepatitis (NASH) are very common in the Western world and strongly associated with obesity. No known effective treatment is known. From animal studies, it is known that the compound resveratrol perhaps has the potential to neutralize obesity-induced diseases. Resveratrol is already widely used as a food supplement though the precise effects are unknown. This project focuses on the effect of Resveratrol on fatty liver disease. The researchers plan to investigate the effects of Resveratrol or placebo treatment for 6 months on NAFLD/NASH in obese patients.

DETAILED DESCRIPTION:
Obesity is associated with non-alcoholic fatty liver disease (NAFLD) and steatohepatitis (NASH) and recently, low-grade inflammation has been hypothesized to be the causative link. From animal studies, it is known that the compound resveratrol (RES) has strong anti-inflammatory and antioxidant effects and perhaps the potential to neutralize obesity-induced diseases. RES is already widely used as a food supplement though the precise effects are unknown. This project focuses on the effect of RES on fatty liver disease. In a double-blind controlled clinical trial, the researchers investigate the effects of RES 500 mg or placebo treatment x 3 daily for 6 months on NAFLD/NASH in 48 obese patients in a double-blind, randomised, controlled clinical trial. The researchers hypothesize that RES improves the ALT levels and reduces liver fat and inflammation assessed by MR spectroscopy and histological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* ALT ≥70 U/L for men and ≥45 U/L for women
* steatosis of the liver, assessed by ultrasonography
* one of the following:

  * waist circumference ≥102 cm for men and ≥88 for women
  * hypertension: BP ≥130/80 mmHg
  * raised triglycerides ≥1,7 mmol/L
  * reduced HDL cholesterol ≤1.0 mmol/L
* BMI ≥ 25 kg/m²

Exclusion Criteria:

* weight > 130 kg
* comorbidity such as diabetes, cancer, metabolic or coagulation disorder, or significant liver-, heart- or kidney disease
* MRI contraindication
* treatment with glucocorticoids or methotrexate
* alcohol intake >20g/daily for men and >12 for women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in hepatic steatosis and inflammation | 6 months
  Changes in hepatic and inflammatory markers ind the blood such as ALT, hs-CRP, TNFa Changes in hepatic fat content, assessed by MR spectroscopy Changes in hepatic steatosis and inflammation, assessed histologically Changes in the expression of proteins in the relevant inflammatory pathways, assessed by gene expression studies

SECONDARY OUTCOMES:
Assessment of tolerability and side-effects | 6 months
  Assessment of tolerability and side-effects of Resveratrol versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, MD, PhD, Principal Investigator — Department of Hepatology and Gastroentology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Dept. of Hepatology and Gastroentology, Aarhus, Denmark